CLINICAL TRIAL: NCT07189208
Title: Evaluation of Antimicrobial Prophylaxis to Prevent Syphilis in Pregnancy in Patients at Risk in Rio de Janeiro, Brazil
Acronym: PRESERvE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Karin Nielsen, Professor of Clinical, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-001337; R01AI187414 (NIH)
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Congenital Syphilis
Keywords: congenital syphilis
MeSH Terms: conditions — Syphilis, Congenital | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Counseling and intensified testing and, if negative, Benzathine Penicillin G (Experimental): Counseling about prevention of STIs at each pre-natal visit. Treponemal and non-treponemal tests every four weeks beginning at the 28th week of pregnancy and at delivery. If negative, IM injection of 2.4 million units of Benzathine Penicillin G. If positive, syphilis treatment based on the guidelines of the Brazilian Ministry of Health.
  Interventions: Drug: Benzathine penicillin 2.4 million units; Behavioral: Counseling and intensified testing.
- Counseling and intensified testing without using Benzathine Penicillin G (Active Comparator): Counseling about prevention of STIs at each pre-natal visit. Treponemal and non-treponemal tests every four weeks beginning at the 28th week of pregnancy and at delivery. If positive, syphilis treatment based on the guidelines of the Brazilian Ministry of Health.
  Interventions: Behavioral: Counseling and intensified testing.

INTERVENTIONS:
Drug: Benzathine penicillin 2.4 million units — IM injection of BPG
  Arms: Counseling and intensified testing and, if negative, Benzathine Penicillin G
Behavioral: Counseling and intensified testing. — Brazilian Ministry of Health guidelines for the prevention and diagnosis of maternal syphilis consist of counseling about STI prevention and syphilis testing at the first pre-natal consultation, at a subsequent consultation during or after 28 weeks of pregnancy, at delivery, and in case of abortion or stillbirth. In this study, intensified testing refers to treponemal and non-treponemal tests once every four weeks beginning as of the 28th week of pregnancy.

SUMMARY:
The goal of this clinical trial is to learn if benzathine penicillin works to prevent maternal syphilis. It will also learn about the safety of benzathine penicillin. The main questions it aims to answer are:

* Does benzathine penicillin lower the rate of syphilis in pregnancy?
* What medical problems do participants have when taking benzathine penicillin? Researchers will compare benzathine penicillin to routine care to see if benzathine penicillin works to prevent syphilis.

Participants will:

* Take benzathine penicillin or receive routine care during the third trimester of pregnancy
* Visit the clinic once a month for injections and tests
* Report any reactions to benzathine penicillin to the study team

DETAILED DESCRIPTION:
Syphilis rates during pregnancy have been rising consistently in Brazil in the last decade, with a parallel increase in the rates of congenital syphilis. The state of Rio de Janeiro, in particular, has consistently had the highest rate of gestational syphilis in the country. It is critical to develop an intervention to reduce the risk of syphilis infection during pregnancy, especially for women most at risk of acquiring congenital syphilis. The investigators hypothesize that routine counseling on prevention of sexually transmitted infections (STIs) and the use of benzathine penicillin G (BPG) prophylaxis during pregnancy may help reduce the rates of syphilis in high risk pregnant populations and congenital syphilis. The investigators propose a randomized, unblinded clinical trial using BPG prophylaxis in pregnant women at higher risk of syphilis during pregnancy. The primary objective is to prevent the development of gestational syphilis and congenital syphilis through counseling on prevention of STIs, monthly treponemal and non-treponemal tests beginning in the 28th week of pregnancy and for those testing negative monthly IM injections of BPG, compared to counseling on prevention of STIs and monthly treponemal and non-treponemal tests beginning in the 28th week of pregnancy (enhanced standard of care). The primary maternal endpoint is a negative POC treponemal test and VDRL test at delivery confirming absence of maternal syphilis infection. The primary infant endpoint is absence of congenital syphilis.

The study population is pregnant persons testing negative for syphilis at 28 weeks' of pregnancy but who are at higher risk of contracting syphilis during pregnancy. The study plans to enroll at the Hospital Federal dos Servidores do Estado or at maternity hospitals. Study participants with a viable pregnancy and no significant pregnancy complications until the time of enrollment who meet the inclusion and exclusion criteria are randomized to receive counseling about prevention of STIs, enhanced serological screening, and if testing negative receive 2.4 million units of BPG IM at 28 weeks of pregnancy (+/- one week), 32 weeks (+/- one week) and 36 weeks (+/- one week) or counseling and enhanced serological screening (enhanced standard of care). The duration of the study will be 3.5 years for recruitment of participants, 6 months to complete follow-up and one additional year for data analysis, data write up and publishing of results. The duration of participation for each pregnant person will be 4 to 5 months (from 28 weeks of gestational age to delivery). Infants will be followed in the neonatal period (first 4 weeks of life).

ELIGIBILITY:
Inclusion Criteria:

1. Uncomplicated, viable pregnancy
2. Elevated risk for syphilis acquisition (one or more of the following):

   1. Prior history of STIs last 3 years
   2. HIV infection
   3. Age < 21 years
   4. In a sexual partnership of < 3 mo., or > 3 sexual partners in the last 6 mo.
   5. Late initiation of prenatal care (> 14 weeks of pregnancy)
   6. Residence in area where syphilis prevalence is 10% or higher.
3. Ability to provide written informed consent
4. No allergy to penicillin
5. Prenatal care at one of the sites participating in the study
6. Ongoing sexual activity during study period.
7. Negative rapid treponemal test at baseline.

Exclusion Criteria:

1. Non-viable pregnancy
2. Very high risk pregnancy
3. Inability to provide written informed consent
4. Allergy to penicillin
5. Positive rapid treponemal test at baseline
6. Lack of sexual activity during study period.
7. Any persisting coagulation disorder that would contraindicate IM injections.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with absence of maternal syphilis infection | Labor and delivery
  Negative POC treponemal test and VDRL test following entry into the study and at the time of labor and delivery confirming absence of maternal syphilis infection. A participant developing a positive serologic result after study entry will have reached a study endpoint and will be followed off study.

SECONDARY OUTCOMES:
Number of participants who agree to the intervention and continue on the regimen after the first visit | First study visit through 28 days after delivery
  For acceptability, the investigators will monitor our recruitment attempts prior to study entry to evaluate how many potential participants were offered study enrollment. For participants who enroll in the study, the investigators will evaluate how many agree to the intervention and continue on the regimen after the first visit, noting any premature study discontinuation and the reason for discontinuation using a questionnaire.
Degree of pain at the injection site from 0 to 10 according to the Numeric Ranking Scale | First study visit through 28 days after delivery
  To assess tolerability, the investigators will offer participants an online questionnaire where they record their experience with the use of IM penicillin during the study, assessing their experience with treponemal and nontreponemal tests (both arms), the degree of pain at the injection site (0 to 10) according to the Numeric Ranking Scale in which higher scores mean worse pain, any local or systemic symptoms afterwards, duration of discomfort, or any other local or systemic findings for each study visit. The investigators will also administer a tolerability questionnaire to participants randomized to the enhanced standard of care.
Number of participants with any cardiovascular adverse event following injection of Benzathine Penicillin G | First study visit to labor and delivery
  Cardiovascular adverse events are defined as any of following: hypotension, palpitations, syncope, tachycardia, and hypersensitivity reactions.
Number of participants with any pregnancy complications | Delivery through 4 weeks after delivery
  Pregnancy complications are defined as emergency C-section or still birth.
Number of participants with any dermatologic adverse event following injection of Benzathine Penicillin G | First study visit to labor and delivery
  A dermatologic adverse event will be defined as any of the following: acute, generalized rash, diaphoresis, dermatitis, infection of skin or other subcutaneous tissues, pruritus, skin discoloration, ulceration at injection site, any type of allergic reaction, or urticaria.
Number of participants with fever following injection of Benzathine Penicillin G | First study visit to labor and delivery
  Fever will be defined as axillary temperature of 37.2°C or higher or rectal, oral, tympanic, or temporal artery temperature of 38°C higher.
Number of participants with any gastrointestinal adverse events following injection with Benzathine Penicillin G | First study visit to labor and delivery
  A gastrointestinal adverse event will be defined as any of the following: hematochezia, nausea, diarrhea, or vomiting
Number of participants with genitourinary adverse events following injection with Benzathine Penicillin G | First study visit to labor and delivery
  A genitourinary adverse event is defined as hematuria or proteinuria.
Number of participants with hepatic adverse events following injection with Benzathine Penicillin G | First study visit to labor and delivery
  A hepatic adverse event is defined as increased transaminases (AST/ALT).
Number of participants with immunologic adverse events following injection with Benzathine Penicillin G | First study visit to labor and delivery
  An immunologic adverse event is defined as eosinophilia or other systemic allergic reactions
Number of participants with local injection site reactions following injection of Benzathine penicillin G | First study visit to labor and delivery
  Local injection site reactions are defined as discomort or aching at the injection site, pain upon touch of the injection site, erythema, swelling, induration, pruritus, or bruising.
Number of participants with neurologic adverse events following injection of Benzathine Penicillin G | First study visit to labor and delivery
  Neurologic adverse events are defined as anxiety, confusion, fatigue, headache, or pain
Gestational age at delivery of live born neonates | Delivery to 28 days after delivery
  Gestational age will be defined based on obstetric ultrasound, date of last menstrual period, or clinical exam at delivery (Capurro method).
Birth weight at delivery of liveborn neonates | Delivery to 28 days after delivery
  Weight in grams
Number of neonates with any neonatal complications | Delivery to 28 days after delivery
  Neonatal complications are defined as neonatal death, low birth weight (<2,500 g), preterm delivery (<37 weeks), or small for gestational age.
Number of neonates admitted to the intensive care unit (ICU) | Delivery to 28 days after delivery
  Number of neonates admitted to the intensive care unit (ICU)
Number of pregnant participants admitted to the hospital for any reason after delivery | Delivery to 28 days after delivery
  Number of pregnant participants admitted to the hospital for any reason after delivery
Number of pregnant participants admitted to the hospital due to delivery complications | Delivery to 28 days after delivery.
  Delivery complications are defined as postpartum hemorrhage, sepsis, perineal tears, or thromboembolism.
Number of pregnant participants with a prolonged hospital stay following delivery | Delivery to 28 days after delivery
  A prolonged hospital stay is defined as more than 72 hours after delivery

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Centro de Referencia e Atenção Especializada a Saúde da Mulher (CRAESM), Duque de Caxias, Rio de Janeiro
  - Policlínica Hospital Municipal Duque de Caxias, Duque de Caxias, Rio de Janeiro
  - Unidade Básica de Saúde José de Freitas, Duque de Caxias, Rio de Janeiro
  - Hospital Federal dos Servidores do Estado, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No